CLINICAL TRIAL: NCT01307202
Title: Multiple Doses of Gabapentin and Postoperative Morphine Consumption in Total Knee Arthroplasty
Brief Title: Morphine Consumption in Joint Replacement Patients, With or Without Gabapentin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-215-TKR
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Post Operative Pain; Total Knee Replacement
Keywords: knee; arthroplasty; postoperative pain; gabapentin
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin 600 mg will be given per oral two hours preoperatively and 200 mg three times daily after surgery (600 mg/day).
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo will match the the gabapentin pill and will be given orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — 600mg of Gabapentin will be given orally preoperatively and 200mg for 3 times a day after surgery for 3 days
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Placebo will match the the gabapentin pill and will be given orally.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Total knee arthroplasty is amongst the most painful procedures postoperatively, and pain management can be a challenge. Different measures have been introduced to manage severe postoperative pain int hese patients. Previous studies have investigated gabapentin in acute postoperative pain and demonstrated reducted pain, postoperative morphine consumption, morphine related side effects, and postoperative pain scores. To date, this analgesia adjunct has yet to be investigated in total joint arthroplasty patients.

DETAILED DESCRIPTION:
The study was submitted to Health Canada and received the letter of no objection. A randomized, double-blind, placebo-controlled study. The randomization scheme will be prepared and will be done by the pharmacy department at McMaster University. Ninety patients undergoing primary knee arthroplasty will be recruited from the preoperative clinic. Forty-five patients in each population will be allocated to a gabapentin group and the other forty-five to a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 19-90
* elective single joint, primary total knee arthroplasty
* use of PCA with morphine for postoperative pain control has been discussed and agreed upon between patient and anesthetist

Exclusion Criteria:

* bilateral total knee arthroplasty
* revision knee arthroplasty
* underlying disease of epilepsy, seizure, or chronic pain syndrome
* active gastrointestinal bleeding within the last 6 months
* history of non-steroidal anti-inflammatory drug (NSAID) induced asthma
* known or suspected history of drug or alcohol abuse
* participant currently takes gabapentin or pregabalin for any reason
* participant currently takes pain medication that is more potency than codeine or oxycodone (morphine, hydromorphone, meperidine, methadone, fentanyl, including any long acting narcotics)
* known allergy to study medications: gabapentin, morphine, NSAID, acetaminophen
* unable to tolerate morphine
* liver impairments
* kidney impairment or calculated creatinine clearance by Cockcroft-Gault formula is <=60ml/min
* pregnancy or breast-feeding
* participant currently receives associated worker's compensation benefits (WSIB)
* participant unable or unwilling to give written or informed consent
* unable to use PCA

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Amount of morphine consumption | 2 years

SECONDARY OUTCOMES:
Side effects | 2 years
  Nausea/Vomiting Sedation Pruritis Visual Disturbance Dizziness/Lightheadness

CONTACTS AND LOCATIONS:
Overall Officials: Manyat Nantha-Aree, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Paul JE, Nantha-Aree M, Buckley N, Shahzad U, Cheng J, Thabane L, Tidy A, DeBeer J, Winemaker M, Wismer D, Punthakee D, Avram V. Randomized controlled trial of gabapentin as an adjunct to perioperative analgesia in total hip arthroplasty patients. Can J Anaesth. 2015 May;62(5):476-84. doi: 10.1007/s12630-014-0310-y. Epub 2015 Mar 14. PMID 25772701
- [Derived] Paul JE, Nantha-Aree M, Buckley N, Cheng J, Thabane L, Tidy A, DeBeer J, Winemaker M, Wismer D, Punthakee D, Avram V. Gabapentin does not improve multimodal analgesia outcomes for total knee arthroplasty: a randomized controlled trial. Can J Anaesth. 2013 May;60(5):423-31. doi: 10.1007/s12630-013-9902-1. Epub 2013 Mar 12. PMID 23479393